CLINICAL TRIAL: NCT02428062
Title: Effect of Target Intraoperative Blood Pressure on the Incidence of Post-operative Cognitive Dysfunction in Patients Aged 75 and Older Undergoing General Anesthesia for Non-cardiac Surgery: an International Multicenter Randomized Controlled Trial
Brief Title: Target Hemodynamics and Brain Injury During General Anesthesia in the Elderly
Acronym: THE BRIDGE
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Pending Pilot study results evaluation
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TB-POCD
Record Dates: First submitted 2015-04-08; First posted 2015-04-28 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Post-operative Cognitive Dysfunction
Keywords: Post-operative complications; Mild cognitive impairment; Delirium
MeSH Terms: conditions — Cognitive Dysfunction; Delirium | interventions — Phenylephrine; Ephedrine; Epinephrine; Norepinephrine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard-of-Care (No Intervention): The intraoperative hemodynamic management of the patients assigned to this arm will be left to the discretion of the anesthesiologist, without any indication as to the intraoperative hemodynamic strategy to be adopted.
- Treatment (Experimental): The anesthesiologist will have as hemodynamic target for patients assigned to this arm the maintenance of mean arterial blood pressure within 10% of the baseline blood pressure value (recorded at the preoperative evaluation). The strategy to reach this hemodynamic target will be left to the clinical judgment of the anaesthesiologist in charge. The possible strategies include a vasoconstrictor agent (either phenylephrine, ephedrine, epinephrine, norepinephrine or dopamine), intravenous fluids, patient's positioning or reduction of depth of anesthesia.
  Interventions: Procedure: Hemodynamic target; Drug: Phenylephrine; Drug: Intravenous fluids; Procedure: Patient's positioning; Procedure: Reduction of depth of anesthesia; Drug: Ephedrine; Drug: Epinephrine; Drug: Norepinephrine; Drug: Dopamine
- Control (No Intervention): Subjects assigned to this arm will undergo the same geriatric, neuropsychologic and audiologic evaluations administered to patients of the "Standard-of-Care" and "Treatment" arms at the same time points (baseline, 3 months and 1 year). These subjects will not undergo any surgical procedure and will therefore not be evaluated for post-operative complications or delirium occurrence.

INTERVENTIONS:
Procedure: Hemodynamic target — The anaesthesiologist is requested to maintain intraoperative mean arterial blood pressure of the patient within 10% of the baseline mean arterial blood pressure (recorded during the preoperative evaluation) of that patient. In order to reach this hemodynamic target the anesthesiologist can choose between one or more of the following four sub-interventions:
  1. vasoconstrictor agents (either phenylephrine, ephedrine, epinephrine, norepinephrine or dopamine)
  2. intravenous fluids
  3. patient's positioning
  4. reduction of depth of anesthesia
  Arms: Treatment
Drug: Phenylephrine — Phenylephrine 0.1-0.2 mg intravenous bolus
  Other Names: Sub-intervention 1: Vasoconstrictor agent
  Arms: Treatment
Drug: Intravenous fluids — A crystalloid fluid bolus is given intravenously (5-10 ml/kg)
  Other Names: Sub-intervention 2
  Arms: Treatment
Procedure: Patient's positioning — The operating table is positioned so that the patient's head lies below the level of the patient's feet (Trendelenburg position) in order to increase venous return
  Other Names: Sub-intervention 3
  Arms: Treatment
Procedure: Reduction of depth of anesthesia — The halogenated anesthetic vapor's inspiratory fraction is decreased in order to reduce the associated peripheral vasodilation
  Other Names: Sub-intervention 4
  Arms: Treatment
Drug: Ephedrine — Ephedrine 5-25 mg intravenous bolus
  Other Names: Sub-intervention 1: Vasoconstrictor agent
  Arms: Treatment
Drug: Epinephrine — Epinephrine 5-10 mcg intravenous bolus
  Other Names: Sub-intervention 1: Vasoconstrictor agent
  Arms: Treatment
Drug: Norepinephrine — Norepinephrine 0.01 - 0.1 mcg/kg/min intravenous continuous infusion
  Other Names: Sub-intervention 1: Vasoconstrictor agent
  Arms: Treatment
Drug: Dopamine — Dopamine 5 - 10 mcg/kg/min intravenous continuous infusion
  Other Names: Sub-intervention 1: Vasoconstrictor agent
  Arms: Treatment

SUMMARY:
BACKGROUND: Post-operative cognitive dysfunction (POCD) is a potentially irreversible loss of brain functions observed in elderly patients after surgical operations under general anaesthesia. POCD at 3 post-operative months is observed in up to 15% of patients aged 70 years and more, and the only recognized risk factor for this condition is increasing age. Importantly, the incidence of POCD at 3 months has been associated to an increased disability and mortality.

OBJECTIVES: The present study will evaluate in patients aged 75 years and older undergoing general anaesthesia for non-cardiac surgery, whether an hemodynamic strategy, aiming at maintaining intra-operative arterial blood pressure close to patient's preoperative blood pressure, i.e., to avoid hypotensive episodes, reduces the incidence of POCD at three months.

METHODS: Around 1800 consecutive patients scheduled to undergo general anaesthesia for elective non-cardiac surgery will be enrolled. Each patient's cognitive function will be evaluated preoperatively and at 3 months and 1 year postoperatively, together with the occurrence of hearing loss and vestibular function impairment. Furthermore, the incidence of postoperative delirium and cardiovascular, respiratory and infectious complications will be evaluated.

EXPECTED RESULTS: The primary outcome is a 25% relative reduction in the incidence of POCD at 3 postoperative months. Secondary outcomes are the reduction of POCD incidence at 1 postoperative year, a reduction in postoperative hearing loss and vestibular impairment at 3 months, a reduction in the incidence of delirium. Hospital length of stay and 90 day mortality will also be assessed. This present study could have a high socio-economic impact, reduce healthcare costs and patient morbidity and mortality with a simple not expensive intraoperative intervention.

DETAILED DESCRIPTION:
BACKGROUND Post-operative cognitive dysfunction (POCD) is defined as a spectrum of postoperative central nervous system dysfunctions both acute and persistent, including subtle neurologic signs and neuropsychological impairment. The incidence of POCD is clearly associated with the age of patients, with older patients being more susceptible to neurologic impairment following anesthesia and surgery. Due to the increasing life expectances and ameliorated surgical and anesthesiologic techniques, more and more elderly people are undergoing surgical procedures. In this respect, POCD is a complication that needs to be taken into account in the perioperative course of elderly patients, especially in those with reduced neurological functional reserve capacity and high prevalence of comorbidities. It is worth underlining that the occurrence of POCD brings a very important subjective burden on the quality of life of the patient and also and outstanding social impact.

Several observational studies have shown that POCD occurs in 25% of patients 1 week after the surgical procedure (early POCD) and in approximately 15% of patients at 3 months (late POCD). Importantly, the incidence of POCD at 3 months has been associated to an increased disability and mortality.

Post-operative cognitive dysfunction is probably a multifactorial syndrome, nevertheless 3 principal pathophysiological hypothesis, that certainly could co-exist, have been formulated:

1. Pharmacological hypothesis: drugs employed during anesthesia can produce alterations in the neuronal network, principally through alterations of the cholinergic transduction signal;
2. Toxic hypothesis: the neuronal damage is a direct consequence of the drugs employed during anesthesia and of the inflammatory mediators associated to the surgical procedure;
3. Hemodynamic hypothesis: hemodynamic changes induced by general anesthesia cause alterations in cerebral blood flow, potentially resulting in ischemic neuronal damage.

The present study focuses on the third hypothesis and aims to evaluate the influence of a target of intraoperative arterial blood pressure based on preoperative values on the development of POCD at 3 months after elective non-cardiac surgery under general anesthesia in patients aged 75 years and older.

The present study has a potential high scientific and socio-economic impact as it could identify a single and quite easily accomplished intraoperative intervention, i.e. a different management of intraoperative blood pressure, that could potentially reduce the incidence of neurological deterioration in elderly patients undergoing general anesthesia for non-cardiac surgery.

Furthermore, it will be the first study investigating a population of patients aged 75 years and more and, to the best of the investigators' knowledge, the first study that will evaluate systematically the possible changes in hearing and vestibular function induced by general anesthesia and surgery.

DETAILED RESEARCH PROTOCOL

The present study is structured in 3 distinct phases:

1. Preoperative Phase;
2. Intraoperative Phase;
3. Postoperative Phase;

1) PREOPERATIVE PHASE After obtaining informed consent to the study, several evaluations are performed in the Clinic for preoperative anesthesiology evaluation. These include the standard anesthesia evaluation, a geriatric and neuropsychological evaluation and an audiology evaluation. All preoperative evaluations are performed on the same day and in the same place during the normal path followed by outpatients scheduled for elective surgery. Geriatric, neuropsychological and audiology evaluation are always performed in the same sequence.

Multidimensional Geriatric Assessment:

The multidimensional geriatric assessment includes several tests that allow a global evaluation of the functional status of the patient, including the cognitive domain and the functional performance (ability).

The Mini Mental State Examination (MMSE) and the Clock Drawing Test will be used to assess the cognitive state of the patients. The MMSE is usually employed in clinical practice for two reasons: (i) as a quick tool to screen the cognitive status of the patient and (ii) as a tool to track the changes over time in cognitive state of the patients. The MMSE consists of 30 items (questions/tests), that explore different cognitive domains: spatial and temporal orientation, memorization of words, attention, calculation, recall, language and constructive praxis. The score of the MMSE ranges therefore from 0 to 30. A corrected score of ≤ 23 is usually considered suggestive of cognitive decline. The score of the MMSE is corrected for age and education of the patient.

The Clock Drawing test (CDT) is an additional test employed to evaluate the global cognitive state of patients and is considered complementary to the MMSE. To perform the CDT the patient is asked to draw a circle in order to symbolize a clock face. Furthermore the patient is asked to draw the watch hands in order to indicate ten past eleven. The test explores the visual-spatial, practical and executive functions of the patient. The maximal obtainable score is 5/5 and requires the presence of all numbers, drawn in the correct order and close to the border of the clock face, with the correct symmetry and the watch hands correctly showing ten past eleven. The presence of extra numbers, segmentation lines or rotation of the numbers determines the subtraction of 1 point to the score. Scores > 3/5 are considered normal.

Functional performance is evaluated employing the scores of the "Activities of Daily Living" (ADL) and the "Instrumental Activities of Daily Living" (IADL), respectively.

The ADL are the activities that a person is able to perform independently on a daily basis (eat, dress, wash themselves, move from bed to the chair, use the toilet, etc.). The IADL are the activities that allow a person to live independently in a house or apartment (cook, clean up the house, take medications, use the phone, etc. ).

Finally the patients will be characterized in terms of frailty. The geriatric concept of frailty generically indicates a condition of increased vulnerability to stressful conditions, associated to an increased risk of adverse events including falls to the ground, disability, hospitalization and mortality. Physical frailty is defined by the presence of 3 or more of the following criteria:

1. Unintentional weight loss (≥ than 5% body weight loss in the last year);
2. General feeling of exhaustion (subjective, based on questions on the effort in performing certain activities);
3. Weakness as expressed by a reduced handgrip strength, applying different reference values for women and men;
4. Slow walking speed;
5. Low levels of physical activity; The presence of 1 or 2 of these criteria characterizes the so called "pre-frailty", a condition that is more sensitive to eventual interventions as compared to frailty (3 or more criteria).

Finally, patients will be evaluated for "cognitive frailty", which combines physical frailty with the score of the Clinical Dementia Rating (CDR) (see below), in order to identify non-dement patients in whom physical frailty is however associated to an initial cognitive impairment.

Patients are classified in 4 different categories:

1. Healthy elderly subjects (no evidence of physical frailty and CDR = 0);
2. Elderly subjects with physical frailty and normal cognitive function (presence of physical frailty and CDR =0);
3. Elderly subjects without physical frailty but with initial cognitive impairment (no physical frailty and CDR = 0.5);
4. Elderly subjects with physical frailty and initial cognitive impairment (presence of physical frailty and CDR = 0.5); The condition of the subjects belonging to group 4 is defined as "cognitive frailty".

The Clinical Dementia Rating (CDR) is a complex scale performed to quantify the severity of the symptoms of dementia. It includes queries about the cognitive and functional domains. The final score ranges between 0 and 3, with higher scores indicating more severe dementia symptoms. A score of 0.5 is suggestive of the presence of mild symptoms. It is therefore possible that patients with corrected MMSE ≥ 24 have a CDR score of 0.5. Of note, patients included in the study will not undergo the CDR test, as the different items that compose the CDR can be derived from the performed geriatric and neuropsychological test batteries (see below).

Neuropsychological Evaluation The cognitive functionality at baseline and its possible worsening after anesthesia/surgery, i.e. the development of POCD, is best evaluated through the administration of neuropsychological test batteries. During the baseline evaluation a neuropsychologist will administer to the patient (or to the subject in the Control group) a battery of tests standardized to evaluate specifically different cognitive domains: memory, attention, language, executive functions, speed of information processing. The obtained raw scores will be corrected for age, gender and education and transformed, according to Italian calibration standards, in standardized scores (Equivalent Scores = ES) on an ordinal scale that ranges from 0 to 4, where 0 represents scores below the cut-off, i.e., pathological scores, 1 that represents borderline scores and 2,3 and 4 which characterize normality.

The duration of the administration of the test battery is approximately 35 minutes. At 3 months and 1 year from the surgical procedure/general anesthesia (or from baseline evaluation in the Control group) the same test battery will be repeated. In those tests having a parallel version, the parallel version will be administered, in order to reduce the learning effect. The difference in scores of the tests performed at 3 months (and 1 year) and baseline, corrected for the mean difference observed in the Control group in the same timeframe, will be used in order to define the occurrence of POCD.

Patients in whom the difference (worsening) in the global score at 3 months to the global score at baseline will be greater than 2 standard deviations from the expected difference, i.e., the mean difference between the two evaluations (baseline and 3 months) observed in the Control Group, will be diagnosed with POCD. Moreover, changes in raw scores of the different tests will be considered with the purpose of identifying possible changes in specific cognitive domains.

The administered neuropsychological tests will be the following:

* Trail Making Test: evaluates the visual-motor coordination and speed and task-switching skills by assessing someone's ability to follow a simple number sequence (Trails A) and a more complex sequence of alternating numbers and letters (Trails B).
* Stroop test: evaluates selective attention, executive functions, the inhibition of distractions and cognitive flexibility.
* Symbol Digit Modalities Test: evaluates sustained attention, with elements of vigilance and working memory.
* Free and Cued Selective Reminding Test: measures anterograde visual and verbal memory skills.
* Verbal Phonemic Fluency Test: measures the capacity of access to verbal vocabulary and is considered a marker of pre-frontal functionality.
* Denomination test: evaluates the capacity of visual access of vocabulary.

These tests have a score and a cut-off value that allows to categorize the result as normal, i.e., that falls within the average results obtained from a control group of healthy subjects matched for age, gender and education, or pathological, i.e., below this average value.

Audiology Evaluation The audiology evaluation will include the following tests: video oculography, pure tone audiometry, disyllabic speech audiometry and speech audiometry with verbal tasks and motor responses.

Video oculography analyzes the function of the oculomotor system through the study of saccadic eye movements and optokinetic system. It allows to identify an alteration at the level of the brainstem, cerebellum or of both structures.

Saccadic eye movements are rapid, ballistic eye movements, which subserve vision by redirecting the visual axis to a new location, i.e., to direct the fovea onto an object or region of interest that appeared in the periphery of the field of view. Saccadic eye movements represent the majority of eye movements and the control signal of saccadic eye movements is the so-called "retinal error".

Collected parameters during the study of saccadic eye movements include:

Latency: this is the time taken from the appearance of a target to the beginning of a saccade in response to that target; Peak Velocity: this is the highest velocity reached during the saccade. Saccade velocity profiles are usually symmetrical at least for small and medium size saccades. In some conditions while the size of saccades remains reasonably accurate, the saccade velocity is greatly reduced - so-called slowed saccades; Precision: relation between angular displacement of the eye and the displacement of the reference target; The "optokinetic reflex" causes eye movement in response to objects moving in the periphery while the head is stationary and is extremely important for stabilizing the image of visual input on the retina and provides for primary control of this capacity when the head is stationary. It is composed by a slow phase (SP), directed toward the movement of the panorama, and a quick phases (QP) with opposite direction. These movements have similar characteristics to saccadic eye movements.

Collected parameters during the study of optokinetic nystagmus include the slow-phase velocity of optokinetic nystagmus, which is dependent upon the speed of the stimulus, gain, expressing the percentage of the ratio between the speed of the slow phase of nystagmus and the speed of the stimulus, asymmetry, indicating the difference in gain between the two sides.

Pure tone audiometry aims at defining quantitatively and qualitatively the possible occurrence of hearing loss, its entity and site of the lesion. Pure tone audiometry is performed through the aid of an audiometer and headphones. This study is performed to investigate the functionality of the peripheral auditory system.

Finally, disyllabic speech audiometry and speech audiometry with verbal tasks and motor responses will be performed, using controlateral masking (cocktail party noise). These evaluations investigate the comprehension of verbal stimuli and numerically quantify the ability to repeat disyllabic words. It also evaluates the semantic comprehension of phrases and the ability of the subject to follow simple motor commands.

These tests, taken together, evaluate both the functionality of the peripheral hearing apparatus and the cortical integration of peripheral signals. Considered parameters are the comprehension of the verbal message (100% represents full understanding) and the sound intensity level at which comprehension is maximal, expressed in decibels hearing level (dB HL). Another parameter studied during speech audiometry testing is the percent reduction of disyllabic words understood as the sound intensity increases. This phenomenon, the reduction of understood disyllabic words with increasing sound intensity, is due to pathologic distortion of cochlear and retro cochlear structures (VIII cranial nerve).

Anesthesiology Evaluation The anesthesiology evaluation will be performed as standard clinical practice in preparation for surgical procedures under general anesthesia. This evaluation will include: physiologic, pathologic and drug history collection, clinical examination including peripheral saturation of oxygen by pulse-oximetry (SpO2), resting heart rate and non-invasive blood pressure measurement with an automatic sphygmomanometer. Three measurements of resting blood pressure will be performed during the visit and the mean value of the three measurements of mean blood pressure will represent the baseline mean arterial blood pressure of the patient

2) INTRAOPERATIVE PHASE. The day of the operation the patient will be randomized to one of two groups, Treatment or Standard of Care (see below). Vital functions will be recorded once the patient is in the operating room, before induction of anesthesia, and throughout the entire duration of the surgical procedure and anesthesia up to extubation or transport to the post-operative intensive care unit. Parameters recorded will include blood pressure (either invasive or non-invasive, depending on clinical need), heart rate, peripheral saturation of oxygen, end-tidal concentration of carbon dioxide, ventilator parameters, drugs and fluid administered, fluid balance and blood loss. Additional measurements will be performed when available: non-invasive cardiac output (Nexfin/Pulsioflex, Edwards Lifesciences), non-invasive cerebral oximetry through near-infrared spectroscopy (INVOS, Covidien) and depth of anesthesia through bispectral index (BIS) measurement (Bispectral Index Technology, Covidien).

The anesthesiologist will be responsible for the clinical management of the patients assigned to the two arms. Violations of the protocol are possible whenever the anesthesiologist judges it clinically necessary.

* Standard of Care Group: intraoperative hemodynamic management will be left to the discretion of the anesthesiologist, without any indication as to the intraoperative hemodynamic strategy to be adopted. Of note, baseline mean arterial pressure (as measured during the preoperative evaluation) will not be communicated to the anesthesiologist in care.
* Treatment Group: in this group the anesthesiologist will have as hemodynamic target the maintenance of mean arterial blood pressure within 10% of the baseline mean arterial blood pressure value. The modalities to reach this target (quantity and type of drugs, quantity and type of intravenous fluids, positioning of the patient etc.) will be left to the clinical judgment of the anaesthesiologist. All interventions will be recorded.

The intraoperative protocol requires the acquisition of hemodynamic, respiratory, and all the other parameters already described at pre-defined intervals (anesthesia induction, start of surgery, every 30 minutes thereafter, end of surgery, extubation/transport to post-surgical ICU).

At the end of the operation the blood pressure recording of the entire duration of general anesthesia will be downloaded from the anesthesia monitor and analyzed offline with a dedicated software to quantify exactly the time spent in each category (mild, moderate or severe, see below) of hypotension or hypertension.

Any hypotensive or hypertensive episode will be classified as mild, moderate or severe based on the worst mean arterial blood pressure recorded during the episode, according to the following cut-offs.

Mild: mean arterial blood pressure 10-20% of baseline mean arterial pressure; Moderate: mean arterial blood pressure 20-40% of baseline mean arterial pressure; Severe: mean arterial blood pressure < or > 40% of baseline mean arterial pressure.

3) POSTOPERATIVE PHASE.

DELIRIUM During the first postoperative week all patients will be evaluated, on a daily basis, for delirium occurrence by the CAM-ICU scale (Confusion Assessment Method for the Intensive Care Unit).

POSTOPERATIVE COMPLICATIONS Length of stay in the ICU (if applicable), length of stay in the hospital and any postoperative complication will be recorded. Cardiac, respiratory, renal, neurologic and hemorrhagic complications will be assessed.

Cardiac complications

Acute myocardial infarction (AMI): detection of a rise and/or fall of cardiac biomarker values (preferably cardiac troponin, cTn) with at least one value above the 99th percentile upper reference limit and with at least one of the following:

* symptoms of ischemia;
* new or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB);
* development of pathological Q waves in the ECG;
* imaging evidence of new loss of viable myocardium or new regional wall motion abnormality;
* identification of an intracoronary thrombus by angiography or autopsy. Congestive heart failure: at least one of the following clinical signs (i.e. elevated jugular venous pressure, respiratory rales/crackles, crepitations, or presence of S3) and at least one of the following radiographic findings (i.e. vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema).

Pulmonary embolism: any one of the following:

1. A high probability ventilation/perfusion lung scan
2. An intraluminal filling defect of segmental or larger artery on a helical CT scan
3. An intraluminal filling defect on pulmonary angiography
4. A positive diagnostic test for deep vein thrombosis (e.g., positive compression ultrasound), acute cor pulmonale at cardiac ultrasound and one of the following:

A. non-diagnostic (i.e., low or intermediate probability) ventilation/perfusion lung scan B. non-diagnostic (i.e., subsegmental defects or technically inadequate study) helical CT scan Cardiac arrest: documented or presumed ventricular fibrillation, sustained ventricular tachycardia, asystole, or pulseless electrical activity requiring cardiopulmonary resuscitation, pharmacological therapy, or cardiac defibrillation.

Atrial fibrillation: new atrial fibrillation that results in angina, congestive heart failure, symptomatic hypotension, or that requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion.

Neurologic complications Stroke (ischemic or hemorrhagic): new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting more than 24 hours or leading to death.

Renal complications Acute kidney injury is defined by an increase in serum creatinine of more than or equal to 1.5 times the baseline (preoperative) value or more than or equal to 0.3 mg/dl.

Hemorrhagic complications Mild hemorrhage: decrease of Hb levels < 3 g/dl without hemodynamic impact, without need for surgical revision or endovascular intervention; conservative treatment (transfusion of 2-3 red blood cells units and fluid infusion); Severe hemorrhage: decrease of Hb levels > 3 g/dl with hemodynamic impact (tachycardia, hypotension, oliguria etc); transfusion of more than 3 red blood cells units; need for surgical revision or endovascular treatment.

POSTOPERATIVE COGNITIVE EVALUATION Patients At 3 months ± 2 weeks and 1 year ± 2 weeks after the surgical intervention, patients will undergo the same geriatric, neuropsychological and audiology evaluations described in the "Preoperative Phase" section.

Subjects of the Control Group Subjects enrolled in the Control group will undergo the same evaluations (geriatric, neuropsychological and audiology) described in the "Preoperative Phase" section and to the same evaluations after 3 months ± 2 weeks and 1 year ± 2 weeks. These subjects will not undergo any surgical procedure and will therefore not be evaluated for post-operative complications or delirium occurrence.

STATISTICS

Sample size calculation.

Primary outcome measure:

The incidence of POCD is around 15% in patients aged over 70 years. Despite the lack of data in patients aged 75 years and more (the average expected age is around 80 years in this population), the investigators estimate an incidence of 20%. Hypothesizing that the proposed intervention (intraoperative arterial blood pressure target) could cause a 25% relative reduction in the incidence of POCD (from 20% to 15%) the sample size, for a probability of type I error α=0.05 and a power (1-β) = 0.8 is of 1812 patients. Of note, at the enrolment of 906 patients the Data Safety and Monitoring Board (DSMB) will perform an ad interim analysis.

Secondary outcome measures:

* Delirium: the incidence of delirium in very old patients undergoing general anesthesia is around 15%. The sample size foreseen for the primary outcome measure (1812 patients) provides a power (1-β) = 0.88 with α = 0.05 to detect a 30% relative reduction in this secondary outcome measure.
* Incidence of POCD at 1 year: the incidence of POCD in patients over 70 years of age, at 1 year after surgery is estimated to be 16%. In the very old, given the lack of data in literature, the investigators estimate that the incidence could be around 20%, therefore similar to the incidence of POCD at 3 months after surgery. The sample size foreseen for the primary outcome measure (1812 patients) provides a power (1-β) = 0.8 with α = 0.05 to detect a 25% relative reduction in this secondary outcome measure.
* Hearing and vestibular dysfunction: There are not sufficient data in the literature to estimate the incidence of this secondary outcome measure. It is therefore not possible to estimate the statistical power.

Design and Pilot Study This is a multicentre international prospective parallel-group double-blind (patients and outcome assessors) randomized controlled trial. Currently two Centres are involved (Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy and Universitätsmedizin Göttingen (UMG), Göttingen, Germany). Other Hospitals will be involved after the enrolment of the first 100 patients (Pilot study).

The first 100 enrolled patients will be included in a formal pilot study in order to evaluate the feasibility of the study and estimate the real incidence of POCD at 3 months in this study population. These patients will be randomized, and the minimization criterion will be applied, similarly to the other patients (see below). Of note, these patients will be included in the final analysis.

Randomization Patients will be randomized on the day of the surgical procedure through the use of a dedicated software.

Considering the known risk factors for POCD (advanced age, major surgery and low level of education), the minimization criterion will be applied to the randomization. Minimization allows to randomize each new patient enrolled in the study in order to minimize the differences between the two allocation arms for the risk factors considered. This means that when a new patient enters the study, the patient's own characteristics for the risk factors considered will affect the patient's probability to be enrolled in one of the two allocation arms. The minimization criterion allows to reduce unbalancing for known risk factors between the allocation arms of the study.

The criteria for minimization will be the following:

* Age class: 75 ≤ age < 80; 80 ≤ age < 85; age ≥ 85
* Foreseen duration of the surgical intervention: < 2 hours; ≥ 2 hours
* Education level (years of scholarity): 0-8 years; 9-13 years; >13 years

Control Group Two hundred and fifty subjects will be enrolled in the Control Group; 30 subjects will be included in the pilot study. Considering the rule of thumb that requires a minimum sample size of 120 for the study of reference intervals, the proposed sample size of 250 seems definitely adequate. Nevertheless, the pilot study will allow to have a clearer view of the application of the parametric method. The sample size of the control group could therefore be resized based on preliminary data from the Pilot Study.

Statistical analysis The analysis of continuous variables will be performed via Student's t-test, one or two way analysis of variance (depending on the characteristics of the analysis). The study of association between continuous variables will be performed through linear regression methods keeping in consideration possible non-linear effects. The analysis of non-categorical variables will be performed with contingency tables through the use of Fisher's exact test and Chi-square test, together with appropriate indicators of association. P<0.05 will be considered as significant. A detailed statistical analysis plan will specify the phases of the analysis in relation to the objectives of the research protocol. Publications deriving from this research protocol will present data according to the current recommendations on parallel-group randomized controlled trials involving non-pharmacological treatments.

The primary and secondary outcomes will be evaluated according an Intention to Treat (ITT) analysis, furthermore results will be evaluated according to the effective adherence to the study protocol ("Per Protocol" Analysis).

Finally, the following pre-specified and subgroups analysis will be performed:

* Total hypotensive time vs. primary and secondary outcome measures;
* Mild, moderate and severe hypotensive time vs. primary and secondary outcome measures;
* Analysis of primary and secondary outcome measures related to minimization categories (age classes, education level, major vs. minor surgery);
* Analysis of primary and secondary outcome measures according to the occurrence of intraoperative cerebral desaturation episodes according to values recorded with the INVOS.
* Analysis of primary and secondary outcome measures in the subgroup of patients with hypertension and in patients with diagnosis of "cognitive frailty".

The study is coordinated by a Steering Committee which includes the scientific representatives of the Institutions assuming all the competences and organizational know-how required for the trial:

Istituto di Anestesia e Rianimazione, Fondazione IRCCS - "Ospedale Maggiore Policlinico, Mangiagalli, Regina Elena", Università degli Studi di Milano [Coordinating Center]: L. Gattinoni, T. Langer, A. Santini, A. Pesenti.

UOC Geriatria, Dipartimento di Medicina Interna e Specializzazioni Mediche,Area di Medicina Interna e Geriatria: D. Mari.

UOC Audiologia, Dipartimento di Medicina Interna e Specializzazioni Mediche, Area di Medicina Specialistica: A. Cesarani Universitaetsmedizin Goettingen, Zentrum Anaesthesiologie-, Rettungs- und Intensivmedizin: M.Quintel.

ELIGIBILITY:
Inclusion Criteria:

* any patient aged 75 years and more scheduled for elective non-cardiac surgery under general anesthesia.

Exclusion criteria:

* Failure to obtain informed consent to the study;
* Impossibility to perform scheduled geriatric and neuropsychological tests during the preoperative evaluation;
* Mini-mental state examination score (corrected for age and education) ≤ 23 at the preoperative evaluation;
* Patients scheduled to undergo intracranic neurosurgical procedures or vascular surgery;
* Patients who have been subjected to a surgical procedure under general anesthesia in the preceding 6 months;
* Patients with metastatic cancer; patients falling in the category of the American Society of Anaesthesiologists (ASA) physical status 4;
* Patients already included in the study, i.e. second surgical procedure;

Inclusion criteria for the Control Group:

• Subjects of 75 years and more in whom no hospitalization or surgical procedure is scheduled in the following 3 months.

Exclusion criteria for the Control Group:

* Failure to obtain informed consent to the study;
* Impossibility to perform scheduled geriatric and neuropsychological tests during the baseline evaluation;
* Mini-mental state examination score (corrected for age and scholarity) ≤ 23 at the baseline evaluation;
* Subjects who have undergone a surgical procedure under general anesthesia in the preceding 6 months;
* Subjects who have undergone an unexpected surgical procedure under general anesthesia in the timeframe between baseline 3 months evaluation.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1812 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative cognitive dysfunction (POCD) at 3 months | 3 months after surgical operation
  For each of the neuropsychological tests a Z-score will be calculated. The Z score represents the magnitude of the deviation (in number of standard deviations) in the test results from the reference (Control Group).
  The Z-score is calculated as the difference between the baseline and the 3 months test result for a patient, corrected for the expected difference (the mean difference for that test observed in the Control Group), divided by the standard deviation of the mean difference for that test observed in the Control Group.
  From the Z-scores of the single tests a combined Z-score can be calculated. Patients in whom the difference (worsening) in the score at 3 months to the score at baseline in at least 2 tests will be greater than 2 standard deviations from the expected difference (i.e. Z-score ≥ 2 in at least 2 tests), will be diagnosed with POCD. Also patients in which the combined Z-score will be equal or greater than 2 will be diagnosed with POCD.

SECONDARY OUTCOMES:
Post-operative cognitive dysfunction (POCD) at 1 year | 1 year after surgical operation
  For each of the neuropsychological tests a Z-score will be calculated. The Z score represents the magnitude of the deviation (in number of standard deviations) in the test results from the reference (Control Group).
  The Z-score is calculated as the difference between the baseline and the 1 year test result for a patient, corrected for the expected difference (the mean difference for that test observed in the Control Group), divided by the standard deviation of the mean difference for that test observed in the Control Group.
  From the Z-scores of the single tests a combined Z-score can be calculated. Patients in whom the difference (worsening) in the score at 1 year to the score at baseline in at least 2 tests will be greater than 2 standard deviations from the expected difference (i.e. Z-score ≥ 2 in at least 2 tests), will be diagnosed with POCD. Also patients in which the combined Z-score will be equal or greater than 2 will be diagnosed with POCD.
Post-operative delirium | Within 7 days after surgical operation
  During the first postoperative week all patients will be evaluated on a daily basis for delirium occurrence by the CAM-ICU scale (Confusion Assessment Method for the ICU).
  The CAM-ICU scale defines delirium by the simultaneous occurrence of items 1, 2 and one between items 3 and 4. Items are listed below:
  1. Acute alteration of mental status or fluctuating mental status in the preceding 24 hours
  2. Inattention
  3. Altered level of consciousness (Richmond Agitation and Sedation Scale, RASS ≠ 0)
  4. Disorganized thinking
Hearing loss at 3 months | 3 months after surgical operation
  Clinical evaluation of worsening in hearing function
Hospital length of stay | Up to 30 days after surgical operation
  Number of days of hospitalization after the surgical operation
Mortality | 90 days
Number of patients with at least one post-operative complication | Within 7 days after surgical operation
  During the first postoperative week patients will be assessed on a daily basis for the occurrence of cardio-pulmonary (acute myocardial infarction, congestive heart failure, pulmonary embolism, cardiac arrest, atrial fibrillation, pneumonia), neurologic (ischemic or hemorrhagic stroke), renal or hemorrhagic complications.
Hearing loss at 1 year | 1 year after surgical operation
  Clinical evaluation of worsening in hearing function
Vestibular dysfunction at 3 months | 3 months after surgical operation
  Clinical evaluation of worsening of vestibular function
Vestibular dysfunction at 1 year | 1 year after surgical operation
  Clinical evaluation of worsening of vestibular function

OTHER OUTCOMES:
Per protocol analysis of outcomes | Up to 30 days after surgical operation, at 3 months and 1 year
  The incidence of the primary and secondary outcomes will be assessed in the Standard of Care arm vs the patients in the Treatment arm who spent at least 75% of the anesthesia time within the hemodynamic target (within 10% of baseline mean arterial blood pressure)
Intraoperative hypotensive times | Up to 30 days after surgical operation, at 3 months and 1 year
  The incidence of the primary and secondary outcomes will be assessed in relation to the absolute and relative time spent in any category of blood pressure defined as "hypotension" (either mild, moderate or severe) and to the absolute and relative time spent in each category of hypotension (mild, moderate or severe). This analysis will be performed on the entire patients population, irrespective of allocation arm.
Intraoperative cerebral desaturations | Up to 30 days after surgical operation, at 3 months and 1 year
  The incidence of the primary and secondary outcomes will be assessed in relation to the absolute and relative time spent with cerebral desaturation (non-invasive cerebral saturimetry < 50%) and to the magnitude of cerebral desaturation episodes. This analysis will be performed on the entire patients population, irrespective of allocation arm.
Subgroup analyses | Up to 30 days after surgical operation, at 3 months and 1 year
  The incidence of the primary and secondary outcomes will be assessed in the following subgroup of patients:
  age stratification categories (age 75-79; 80-84; ≥ 85) surgery stratification categories (minor vs major surgery) education level (<8 years; 8-13 years; > 13 years education) normotensive vs hypertensive patients non-frail patients vs cognitive frail patients

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Gattinoni, MD, FRCP, Principal Investigator — Dipartimento di anestesiologia terapia intensiva e scienze dermatologiche; Thomas Langer, MD, Study Chair — Dipartimento di Anestesia, Rianimazione ed Emergenza Urgenza, Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico, Milano, Italy; Alessandro Santini, MD, Study Chair — Dipartimento di anestesiologia terapia intensiva e scienze dermatologiche; Michael Quintel, MD, PhD, Study Chair — University of Göttingen, Zentrum Anaesthesiologie-, Rettungs- und Intensivmedizin; Antonio Pesenti, MD, Study Chair — Dipartimento di Emergenza Urgenza, Azienda Ospedaliera San Gerardo, Monza,Italy
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico; Via F. Sforza 35, Milan, Italy

REFERENCES:
- [Background] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Background] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706
- [Background] SIMPSON BR, WILLIAMS M, SCOTT JF, SMITH AC. The effects of anesthesia and elective surgery on old people. Lancet. 1961 Oct 21;2(7208):887-93. No abstract available. PMID 13913203
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Abildstrom H, Rasmussen LS, Rentowl P, Hanning CD, Rasmussen H, Kristensen PA, Moller JT. Cognitive dysfunction 1-2 years after non-cardiac surgery in the elderly. ISPOCD group. International Study of Post-Operative Cognitive Dysfunction. Acta Anaesthesiol Scand. 2000 Nov;44(10):1246-51. doi: 10.1034/j.1399-6576.2000.441010.x. PMID 11065205
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Rasmussen LS, Christiansen M, Hansen PB, Moller JT. Do blood levels of neuron-specific enolase and S-100 protein reflect cognitive dysfunction after coronary artery bypass? Acta Anaesthesiol Scand. 1999 May;43(5):495-500. doi: 10.1034/j.1399-6576.1999.430502.x. PMID 10341995
- [Background] Rasmussen LS, Christiansen M, Rasmussen H, Kristensen PA, Moller JT. Do blood concentrations of neurone specific enolase and S-100 beta protein reflect cognitive dysfunction after abdominal surgery?ISPOCD Group. Br J Anaesth. 2000 Feb;84(2):242-4. doi: 10.1093/oxfordjournals.bja.a013410. PMID 10743460
- [Background] Mandal PK, Bhavesh NS, Chauhan VS, Fodale V. NMR investigations of amyloid-beta peptide interactions with propofol at clinically relevant concentrations with and without aqueous halothane solution. J Alzheimers Dis. 2010;21(4):1303-9. doi: 10.3233/jad-2010-100396. PMID 21504123
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840
- [Background] van Beek AH, Claassen JA, Rikkert MG, Jansen RW. Cerebral autoregulation: an overview of current concepts and methodology with special focus on the elderly. J Cereb Blood Flow Metab. 2008 Jun;28(6):1071-85. doi: 10.1038/jcbfm.2008.13. Epub 2008 Mar 19. PMID 18349877
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Shulman KI. Clock-drawing: is it the ideal cognitive screening test? Int J Geriatr Psychiatry. 2000 Jun;15(6):548-61. doi: 10.1002/1099-1166(200006)15:63.0.co;2-u. PMID 10861923
- [Background] Katz S. Assessing self-maintenance: activities of daily living, mobility, and instrumental activities of daily living. J Am Geriatr Soc. 1983 Dec;31(12):721-7. doi: 10.1111/j.1532-5415.1983.tb03391.x. PMID 6418786
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Bohannon RW, Bear-Lehman J, Desrosiers J, Massy-Westropp N, Mathiowetz V. Average grip strength: a meta-analysis of data obtained with a Jamar dynamometer from individuals 75 years or more of age. J Geriatr Phys Ther. 2007;30(1):28-30. PMID 19839178
- [Background] Kelaiditi E, Cesari M, Canevelli M, van Kan GA, Ousset PJ, Gillette-Guyonnet S, Ritz P, Duveau F, Soto ME, Provencher V, Nourhashemi F, Salva A, Robert P, Andrieu S, Rolland Y, Touchon J, Fitten JL, Vellas B; IANA/IAGG. Cognitive frailty: rational and definition from an (I.A.N.A./I.A.G.G.) international consensus group. J Nutr Health Aging. 2013 Sep;17(9):726-34. doi: 10.1007/s12603-013-0367-2. PMID 24154642
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Capitani E, Laiacona M. Composite neuropsychological batteries and demographic correction: standardization based on equivalent scores, with a review of published data. The Italian Group for the Neuropsychological Study of Ageing. J Clin Exp Neuropsychol. 1997 Dec;19(6):795-809. doi: 10.1080/01688639708403761. PMID 9524875
- [Background] Giovagnoli AR, Del Pesce M, Mascheroni S, Simoncelli M, Laiacona M, Capitani E. Trail making test: normative values from 287 normal adult controls. Ital J Neurol Sci. 1996 Aug;17(4):305-9. doi: 10.1007/BF01997792. PMID 8915764
- [Background] Caffarra P, Vezzadini G, Dieci F, Zonato F, Venneri A. Rey-Osterrieth complex figure: normative values in an Italian population sample. Neurol Sci. 2002 Mar;22(6):443-7. doi: 10.1007/s100720200003. PMID 11976975
- [Background] Nocentini U, Giordano A, Di Vincenzo S, Panella M, Pasqualetti P. The Symbol Digit Modalities Test - Oral version: Italian normative data. Funct Neurol. 2006 Apr-Jun;21(2):93-6. PMID 16796824
- [Background] Frasson P, Ghiretti R, Catricala E, Pomati S, Marcone A, Parisi L, Rossini PM, Cappa SF, Mariani C, Vanacore N, Clerici F. Free and Cued Selective Reminding Test: an Italian normative study. Neurol Sci. 2011 Dec;32(6):1057-62. doi: 10.1007/s10072-011-0607-3. Epub 2011 May 19. PMID 21594655
- [Background] Novelli G., Papagno C., Capitani E., Laiacona N., Vallar G., Cappa S.F., Tre test clinici di ricerca e produzione lessicale. Taratura su soggetti normali, Archivio di Psicologia, Neurologia e Psichiatria 1986 oct-dec; vol. 47 (4): 477-506
- [Background] Catricala E, Della Rosa PA, Ginex V, Mussetti Z, Plebani V, Cappa SF. An Italian battery for the assessment of semantic memory disorders. Neurol Sci. 2013 Jun;34(6):985-93. doi: 10.1007/s10072-012-1181-z. Epub 2012 Sep 9. PMID 22960873
- [Background] Audiometria pratica : casi clinici / A. Cesarani ; [a cura di] A. Cesarani. - Torino : Omega Edizioni, 2012. - ISBN 8872415454.
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for Universal Definition of Myocardial Infarction; Authors/Task Force Members Chairpersons; Thygesen K, Alpert JS, White HD; Biomarker Subcommittee; Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA; ECG Subcommittee; Chaitman BR, Clemmensen PM, Johanson P, Hod H; Imaging Subcommittee; Underwood R, Bax JJ, Bonow JJ, Pinto F, Gibbons RJ; Classification Subcommittee; Fox KA, Atar D, Newby LK, Galvani M, Hamm CW; Intervention Subcommittee; Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J; Trials & Registries Subcommittee; Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML; Trials & Registries Subcommittee; Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G; Trials & Registries Subcommittee; Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D; Trials & Registries Subcommittee; Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG); Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S; Document Reviewers; Morais J, Aguiar C, Almahmeed W, Arnar DO, Barili F, Bloch KD, Bolger AF, Botker HE, Bozkurt B, Bugiardini R, Cannon C, de Lemos J, Eberli FR, Escobar E, Hlatky M, James S, Kern KB, Moliterno DJ, Mueller C, Neskovic AN, Pieske BM, Schulman SP, Storey RF, Taubert KA, Vranckx P, Wagner DR. Third universal definition of myocardial infarction. J Am Coll Cardiol. 2012 Oct 16;60(16):1581-98. doi: 10.1016/j.jacc.2012.08.001. Epub 2012 Sep 5. No abstract available. PMID 22958960
- [Background] Devereaux PJ, Sessler DI, Leslie K, Kurz A, Mrkobrada M, Alonso-Coello P, Villar JC, Sigamani A, Biccard BM, Meyhoff CS, Parlow JL, Guyatt G, Robinson A, Garg AX, Rodseth RN, Botto F, Lurati Buse G, Xavier D, Chan MT, Tiboni M, Cook D, Kumar PA, Forget P, Malaga G, Fleischmann E, Amir M, Eikelboom J, Mizera R, Torres D, Wang CY, Vanhelder T, Paniagua P, Berwanger O, Srinathan S, Graham M, Pasin L, Le Manach Y, Gao P, Pogue J, Whitlock R, Lamy A, Kearon C, Chow C, Pettit S, Chrolavicius S, Yusuf S; POISE-2 Investigators. Clonidine in patients undergoing noncardiac surgery. N Engl J Med. 2014 Apr 17;370(16):1504-13. doi: 10.1056/NEJMoa1401106. Epub 2014 Mar 31. PMID 24679061
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Grutzmann R, Ruckert F, Hippe-Davies N, Distler M, Saeger HD. Evaluation of the International Study Group of Pancreatic Surgery definition of post-pancreatectomy hemorrhage in a high-volume center. Surgery. 2012 Apr;151(4):612-20. doi: 10.1016/j.surg.2011.09.039. Epub 2011 Nov 16. PMID 22088819
- [Background] Jennen-Steinmetz C, Wellek S. A new approach to sample size calculation for reference interval studies. Stat Med. 2005 Oct 30;24(20):3199-212. doi: 10.1002/sim.2177. PMID 16189809
- [Background] Moher D, Schulz KF, Altman D; CONSORT Group (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. JAMA. 2001 Apr 18;285(15):1987-91. doi: 10.1001/jama.285.15.1987. PMID 11308435
- [Derived] Langer T, Santini A, Zadek F, Chiodi M, Pugni P, Cordolcini V, Bonanomi B, Rosini F, Marcucci M, Valenza F, Marenghi C, Inglese S, Pesenti A, Gattinoni L. Intraoperative hypotension is not associated with postoperative cognitive dysfunction in elderly patients undergoing general anesthesia for surgery: results of a randomized controlled pilot trial. J Clin Anesth. 2019 Feb;52:111-118. doi: 10.1016/j.jclinane.2018.09.021. Epub 2018 Sep 20. PMID 30243062